CLINICAL TRIAL: NCT05308550
Title: Clinical Evaluation of Rapid RNA Test for Covid-19
Acronym: CERrnaTc-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: West Hertfordshire Hospitals NHS Trust (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 56505; 283408 (Other: IRAS)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two cohorts, the second with a modified version of the test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Other): Version 1 of the rapid test:
  The clinician taking the nasopharyngeal / oropharyngeal swab for standard PCR testing for Covid-19 collected a second swab directly afterwards for the rapid RNA test. The swab was placed in a dry tube, labelled with the patient's ID, date and time of taking the sample, and was taken to the microbiology laboratory for processing.
  In the laboratory, 2ml of RNase-free water was added to the tube and shaken with the swab. Twenty-five microlitres of the swab solution was transferred into a PCR tube containing the dried reagents for the rapid RNA test. This tube was then incubated for 45 minutes at 65'C, then taken out to cool down. The colour of the tube was recorded by the laboratory technician.
  Interventions: Diagnostic Test: rapid RT-LAMP test to detect SARS-COV-2 RNA
- Phase 2 (Other): Version 2 of the rapid test:
  The clinician taking the nasopharyngeal / oropharyngeal swab for standard PCR testing for Covid-19 collected a second swab directly afterwards for the rapid RNA test. The swab was placed in a tube containing 1ml of normal saline (instead of a dry tube). If the patient was eligible but the standard swab had already been taken >12 hours before, we asked them for their consent to take a second standard swab alongside the swab for the rapid RNA test, to ensure that the samples were comparable.
  In the laboratory, the swab was heated to 95'C for 5 minutes to inactivate the virus. Nine ml of RNase-free water was added to the tube and shaken with the swab, before transferring 25ul of the swab solution into the PCR tube containing the dried reagents. This tube was then incubated for 30 minutes at 65'C, then the colour of the tube was recorded and photographed by the laboratory technician at 30 minutes (primary reading) and 45 minutes (secondary reading).
  Interventions: Diagnostic Test: rapid RT-LAMP test to detect SARS-COV-2 RNA

INTERVENTIONS:
Diagnostic Test: rapid RT-LAMP test to detect SARS-COV-2 RNA — rapid RT-LAMP test to detect SARS-COV-2 RNA

SUMMARY:
A new Rapid RNA test for Covid-19 has been developed by Professor Cui and his team at the Department of Engineering Science at the University of Oxford. This can give results in 30 minutes which is much faster than the routine PCR test, which often takes 2-3 days to produce results. In this study we aim to establish the sensitivity of the rapid RNA test, which has never before been evaluated clinically. Preliminary anecdotal evidence suggests that the test is easy to use and appears to give valid results. This initial trial aims to establish whether the sensitivity of this tests is above the threshold of 90%. We aim to include at least 173 patients with symptoms of Covid-19 in Watford General Hospital.

DETAILED DESCRIPTION:
Rapid, accurate diagnosis of Covid-19 would greatly help to improve clinical management of patients presenting with symptoms of possible Covid-19. Currently, results of the standard test for the virus take 2-3 days to be reported. The University of Oxford Institute of Biomedical Engineering has designed a new test, which can produce results in 30 minutes. This uses a nasal/throat swab like the current standard test.

In the first phase of the trial, the swab was sent to the laboratory in a dry tube. In the laboratory, the swab was put into a vial of 1 mL water, and a small amount (25 µL) of the water was put into a test tube. This test tube contained materials which can detect the presence of the novel Coronavirus (SARS-CoV-2). The test tube is then simply warmed to 65°C for 30 minutes, and if the Coronavirus is present, the reagent will change colour from pink to yellow (positive). If there is no virus present in the sample, the colour remains pink (negative). This is designed to be a very simple test that does not need specialist skills or equipment, and so could be carried out in hospitals and even in primary care. In this study we aimed to evaluate the accuracy of this new test. We planned to take a second swab from patients with suspected Covid-19 at Watford General hospital (who were being tested anyway) and to use these swabs to conduct the new test (in ideal laboratory conditions) as well as the standard test. As we were not sure of the accuracy of the new test, its results were not used to make decisions about treatment for the patient. In the initial cohort of 173 patients, Discrepancies were noted with some samples when compared to reference lab results. We then investigated whether the patients who had a positive rapid RNA test, but a negative "gold standard" test, were true positives, by inviting them to have an antibody test. This revealed that 20 of 161 patients with a negative reference test had a false positive result on the rapid test. These false positives may result from interfering substances in the clinical samples, which affect the colorimetric detection based on pH changes.

In view of these first results and feedback, the Oxford team made a number of modifications to the rapid test:

1. Viral inactivation - the swab is placed in saline and heated at 95°C for 5 mins - which kills the virus and makes it safe to use at the point of care
2. The sample is diluted 1 in 10 to avoid interaction with saliva
3. A "molecular switch" was added to avoid false positives.

The diagnostic accuracy of the modified test was then evaluated. We invited patients who were being screened, and patients who had been screened and found to be positive, to take part in this study. As the prevalence of COVID-19 amongst tested patients was lower than we had estimated when calculating the sample size (only 12 of 173 were positive on the reference test), the sample was increased by a further 300 patients. We aimed to discover rapidly whether the modified test is accurate.

The rapid RNA test has the potential to be a useful screening tool if it acquires comparable sensitivity to the current "gold standard" with a rapid and feasible approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting to hospital with symptoms of Covid-19 OR who are asymptomatic but being screened for Covid-19 (including in hospital and drive-through testing centres)
2. Age 18 or over
3. Swab is being taken for standard PCR test of Covid-19
4. Willing and able to give written informed consent

Exclusion Criteria:

1. Lack of written consent
2. Age under 18
3. Routine PCR test not being conducted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity compared to standard PCR | within 12 hours
  Test swab taken within 12 hours of the standard PCR swab

CONTACTS AND LOCATIONS:
Overall Officials: Michael Moore, FRCGP, Principal Investigator — University of Southampton
Locations (1):
- Watford General Hospital, Watford, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No